CLINICAL TRIAL: NCT01840280
Title: Open, Multicenter Observational Study of Irinotecan Utilized in Mono- or Combination Therapy for the Treatment of Advanced Colorectal Carcinoma.
Brief Title: A Non Interventional Study With Irinotecan Onkovis (Irinotecan) Utilized for the Treatment of Cancer
Status: Completed | Type: Observational
Sponsor: Onkovis GmbH (Industry)
Collaborators: AKP Freiburg GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ONKOIRI01
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Carcinoma
Keywords: carcinoma; colorectal cancer; ambulant chemotherapy; treatment cycles; Irinotecan; Irinotecan onkovis; Quantity of Irinotecan; Packaging Sizes
MeSH Terms: conditions — Carcinoma; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carcinoma, Irinotecan onkovis (Irinotecan): Treatment in mono- or combination therapy with Irinotecan of advanced colorectal carcinoma.

SUMMARY:
The main purpose of this observational study with Irinotecan onkovis is to determine the number of treatment cycles and the quantity of Irinotecan onkovis needed for this purpose under the special circumstances of ambulant chemotherapy.

Onkovis aims to contribute to an economical utilization of the chemotherapeutics. This includes provision of appropriate packaging sizes to decrease the excess quantity to be discarded, and thus also follows this objective.

Secondary objective is the assessment of the side effects of Irinotecan onkovis. To this end, data regarding co-medication and adverse events are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Indication for Irinotecan according to the SmPC and treating physician

Exclusion Criteria:

* according to the Irinotecan SmPC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in practices, clinics, hospitals
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The Quantity of Irinotecan onkovis needed per treatment cycle | up to 24 weeks
  Determine the quantity of Irinotecan onkovis needed pro treatment cycle

SECONDARY OUTCOMES:
Adverse events during and after treatment | up to 24 weeks
  The number and kind of adverse events during and after the intra-venous application of Irinotecan will be assessed and documented.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Practice, Elstra
  - Practice, Leipzig
  - Practice, Naunhof
  - Practice, Neustadt/Sachsen
  - Practice, Werdau